CLINICAL TRIAL: NCT05442112
Title: A Randomized Control Trial of eHealth Wellness Behavioral Interventions and Patient-reported Outcomes
Brief Title: Trial of eHealth Wellness Behavioral Interventions and Patient-reported Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00310601
Record Dates: First submitted 2022-06-28; First posted 2022-07-01 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Patients will be randomized 1:1 within provider schedules to either receive a secure message containing a set script on wellness-related topics in MS, or no additional information other than that provided by their clinician.
Who Masked: Participant, Care Provider
Masking Description: Participants will not know which arm they are assigned to, and neither will their provider.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wellness Smartphrase (Experimental): This arm will receive a secure message after the conclusion of their standard clinic visit providing a set script containing information on a number of wellness-related topics in MS (sleep, diet, exercise).
  Interventions: Behavioral: Wellness Patient Message
- No Intervention (No Intervention): This arm will not receive a secure message after their appointment, and will instead receive their standard care with their provider.

INTERVENTIONS:
Behavioral: Wellness Patient Message — The intervention is a detailed patient message containing information on strategies for exercise in MS, how to maintain proper sleep, and dietary improvements to maximize health. These strategies are derived from information provided by the National MS Society in their website and covers these topics in greater detail than would normally be addressed in a normal clinic visit. The message also directs patients to the National MS Society website if they would like more information.
  Arms: Wellness Smartphrase

SUMMARY:
In this project, the investigators hope to evaluate effective methods of communication with patients with multiple sclerosis regarding habits of physical activity, sleep, and diet. Currently, there is weak evidence regarding how to deliver adequate information at scale in the clinics with respect to diet, exercise, and sleep. It is unclear if receiving structured information impacts patient-reported outcomes in multiple sclerosis (MS).

The study team hopes to evaluate the efficacy of after visit direct patient messaging in promoting any behavioral changes, the sustainability of those behavioral changes, and most importantly, if those changes impact patient-reported sense of self-efficacy in the participants disease management. In addition, the study team hopes that the data collected during this study will provide answers on how providing wellness strategies impacts patient reported outcomes, markers of behavior, and sense of disease progression.

DETAILED DESCRIPTION:
This will be a prospective randomized control trial assessing the impact of the delivery of wellness-related information on patient-reported outcomes in multiple sclerosis. The investigators plan to query all patients who meet inclusion criteria over the course of at least three consecutive months who will be seen at the Johns Hopkins Outpatient Center Multiple Sclerosis clinic. On average, 200 patients are seen in the MS clinic monthly, and the investigators hope to enroll 120 patients in this time period. If the investigators are unable to reach this target number in two months, the investigators will continue to message patients over consecutive months until the investigators reach this number. The study team will send a recruitment message through MyChart to all eligible patients prior to the patients next clinic appointment to participate in the study, after which the patients will be consented (with documentation of waiver of consent) if interested. Those who are interested will be asked to fill out a series of electronic baseline questionnaires prior to the patient's appointment (sent by REDCap using subject-specific links).

Participants will subsequently be randomized 1:1 (stratified within each provider's daily clinic schedule) to either receive a secure message providing a set script (see Supplementary Materials) containing information on a number of wellness-related topics in MS (sleep, diet, exercise), or to receiving no additional information other than that provided by the participants clinician. This message will be sent as a secure message through Epic by a member of the study team by the end of the clinic day.

At one month and three months after the clinic visit, the study team will send the same questionnaires as were sent at baseline, assessing self-efficacy, reported physical activity, dietary habits, and sleep quality through REDCap subject-specific links.

The investigators will assess for any differences in outcomes between the control group and the group who received the wellness-related secure message. The investigators will evaluate for covariates that were imbalanced and adjust models when imbalance did occur, which is plausible given the expected sample size. In addition, the investigators will also evaluate via chart review whether diet, exercise, and sleep were assessed or discussed during the clinic visit.

In addition, the investigators will use descriptive statistics to describe participants and compare those who agree versus those who do not agree to participate. The investigators hope to evaluate density of use of the electronic medical record amongst this cohort, as well as demographic data on social determinants of health, including race, socioeconomic status, and geographic location, in order to evaluate predictors of responsiveness to the messaging.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-89 years of age
* Diagnosis of MS (G35) seen at the Johns Hopkins MS Precision Medicine Center of Excellence within the past year, and upcoming appointment within the three-month window. We will require the relevant ICD10 code to be documented at least twice in two separate visits, either in the problem list and/or visit diagnosis, in order to avoid misdiagnosis.
* MyChart active account
* Provides consent to complete questionnaires and undergo randomization

Exclusion Criteria:

* Patients known to be deceased in Epic
* Patients who have opted out of being contacted for research recruitment
* Patients who have opted out of being contacted for MyChart recruitment
* Patients who have opted out of being contacted for any reason

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2023-06-11 (Actual); Primary Completion 2024-05-11 (Actual); Study Completion 2024-05-11 (Actual)

PRIMARY OUTCOMES:
Change in self-efficacy as assessed by the MS Self-Efficacy Scale (MSSE) | Baseline, 1 month, 3 months
  Patients will take the MS Self-Efficacy Scale (MSSE), which has a score range 90-900, with higher scores reflecting greater sense of self-efficacy

SECONDARY OUTCOMES:
Change in Sleep Disturbance the Neuro-Quality of Life Sleep disturbance short form | Baseline, 1 month, 3 months
  Patient-reported outcomes on the Neuro-Quality of Life Sleep disturbance short form, which has a score range of 8-40, with higher scores reflecting better quality of sleep.
Change in Diet behavior Scores as assessed by the Mediterranean-DASH Intervention for Neurodegenerative Delay score (MIND Diet score) | Baseline, 1 month, 3 months
  Patient-reported behaviors on diet through the Mediterranean-DASH Intervention for Neurodegenerative Delay score (MIND Diet score), which has a score range of 0-15, with higher scores reflecting a higher, healthier, quality of diet.
Change in Reported physical activity as assessed by the Godin Leisure-Time Exercise Questionnaire (GLTEQ) | Baseline, 1 month, 3 month
  Patient-reported behaviors on physical activity through the Godin Leisure-Time Exercise Questionnaire (GLTEQ). The score range is from 0-119, with higher scores reflecting a greater degree of physical exercise.
Change in Reported physical activity as assessed by the International Physical Activity Questionnaire (IPAQ) short form | Baseline, 1 month, 3 month
  Patient-reported behaviors on physical activity through the International Physical Activity Questionnaire (IPAQ) short form. Results are reported in metabolic minutes (MET-min), and are continuous, with range of 0-200,000 per week, and higher scores indicating greater physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Shuvro Roy, MD, Study Director — Johns Hopkins University; Ellen Mowry, MD, Principal Investigator — Johns Hopkins University; Scott Newsome, MD, Study Director — Johns Hopkins University; Peter Calabresi, MD, Study Director — Johns Hopkins University; Shiv Saidha, MBBCh, Study Director — Johns Hopkins University; Pavan Bhargava, MD, Study Director — Johns Hopkins University; Michael Kornberg, MD, Study Director — Johns Hopkins University
Locations (1):
- Johns Hopkins Outpatient Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data

REFERENCES:
- [Background] Motl RW, Mowry EM, Ehde DM, LaRocca NG, Smith KE, Costello K, Shinto L, Ng AV, Sullivan AB, Giesser B, McCully KK, Fernhall B, Bishop M, Plow M, Casaccia P, Chiaravalloti ND. Wellness and multiple sclerosis: The National MS Society establishes a Wellness Research Working Group and research priorities. Mult Scler. 2018 Mar;24(3):262-267. doi: 10.1177/1352458516687404. Epub 2017 Jan 12. PMID 28080254
- [Background] Motl RW, McAuley E, Snook EM, Gliottoni RC. Physical activity and quality of life in multiple sclerosis: intermediary roles of disability, fatigue, mood, pain, self-efficacy and social support. Psychol Health Med. 2009 Jan;14(1):111-24. doi: 10.1080/13548500802241902. PMID 19085318